CLINICAL TRIAL: NCT02719730
Title: The Metabolic Impact of Concurrent Food Insecurity and Obesity
Brief Title: Upgrade the Grains Study: Increasing Whole Grain Consumption in Low-income Children With Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in study design to be a pilot with no randomization to intervention/control
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-064
Record Dates: First submitted 2016-03-15; First posted 2016-03-25 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reimbursement arm (Experimental): Participating caregivers will turn in receipts from grocery store purchases. At each of three study visits, participants in the reimbursement arm will receive reimbursement of up to 10% of their usual SNAP benefits for specific whole grain foods purchased at one of two chain stores in the previous month.
  Interventions: Behavioral: Reimbursement for whole grain purchases
- Control arm (No Intervention): Participating caregivers will mail in receipts from grocery store purchases. Participants in the control arm will also be given the same guidance about preferred whole grain foods and whole grain products but will have no specific financial incentive related to purchases of whole grain foods during the 12-week study period.

INTERVENTIONS:
Behavioral: Reimbursement for whole grain purchases — All participants will receive education about whole grain foods. Those in the experimental arm will have a monthly financial incentive for purchases of specific whole grain foods foods during the 12-week study period, whereas the control group will not have a financial incentive for whole grain purchases during the study period.
  Arms: Reimbursement arm

SUMMARY:
This study will assess the impact of a randomized intervention aimed at increasing consumption of whole grain foods among children from low-income households that participate in the Special Nutrition Assistance Program (SNAP, or "food stamps"). A total of 60 obese children (8 to 16 years) will be recruited from a clinical population (Healthy Eating Active Living Program) at University of California San Francisco (UCSF) Benioff Children's Hospital Oakland. Participants and their caregivers will all receive education about whole grain foods, and will be randomized to either an intervention or control group. The intervention group will receive a monthly reimbursement allotment of up to 10% of their usual SNAP benefit for specific whole grain foods purchased during the three month study period. The control group will not have the financial incentive for purchasing whole grain foods during the 12 week study period. The investigators will assess the feasibility of the intervention, the impact of the intervention on household grocery purchases, and the impact on the child's anthropometrics, dietary intake of whole grain foods (24-hour recall), and markers of metabolic risk.

DETAILED DESCRIPTION:
RUN-IN PHASE (Weeks -4 to 0)

* Participants will participate in a "run-in phase" where they will be asked to keep all grocery receipts for a 4 week period

RANDOMIZATION (Week 0)

* Child participants with caregivers who are able to successfully complete the run-in phase are then randomized at that point to be either in the intervention arm or the control arm.
* Patients will be block randomized by age group (8-11 and 12-16).

ACTIVE PHASE (Weeks 0-12)

* Participants will be given education about whole grains and whole grain preparation. Intervention and control participant activities described elsewhere.

RETURN VISIT (Week 24)

* 12 weeks after the completion of the active phase of the study, patients will be asked to return for a final visit at the research center, during which they will also have blood tests and other study activities repeated for one final time.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI greater than 95th percentile for age and gender)
* Low-income family currently participating in SNAP ("food stamps")
* Participant and caregiver speaks either English or Spanish

Exclusion Criteria:

* medications to lower lipid levels (statins), which would affect insulin sensitivity (e.g. metformin, abilify) or which are known to affect serum cholesterol (e.g. carbamazepine).
* Type II diabetes

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2016-08-02 (Actual); Study Completion 2016-08-02 (Actual)

PRIMARY OUTCOMES:
Change in whole grains consumption (ounce equivalents) | Baseline and 3 months
  Using the Nutrition Data System for Research (NDSR) for 24-hour food recall, intake of whole grains (and refined grains, and proportion of grains that are whole) will be assessed. The change in this dietary outcome at the end of 3 months will be evaluated for intervention participants compared to controls.

SECONDARY OUTCOMES:
Change in serum triglycerides (mg/dl) | Baseline and 3 months
  Fasting lipid panel at the end of three month period will be compared to baseline lipid panel: serum triglycerides will be an outcome of particular interest given the intervention.
Change in TG/HDL ratio | Baseline and 3 months
  Fasting lipid panel at the end of three month period will be compared to baseline lipid panel: the ratio of serum triglycerides (TG) to high-density lipoprotein (HDL-C) will be an outcome of particular interest given the intervention.
Change in body mass index (BMI, or kg/m2) | Baseline and 3 months
  The change in BMI after the 3 month intervention period will be examined for intervention group compared to control group.
Change in waist to height ratio (WHtR) | Baseline and 3 months
  Change in waist to height ratio at the end of the 3 month period will be examined for intervention group compared to control group.
Change in proportion of subjects with pre-diabetes | Baseline and 3 months
  The proportion of subjects with prediabetes (using both criteria of Hemoglobin A1c greater than or equal to 5.7% and fasting glucose greater than or equal to 100 mg/dl) after the 3 month intervention period will be compared for intervention and control groups.
Change in percent of monthly SNAP benefit spent on whole grain purchases (dollars) | Baseline and 3 months
  Using collected grocery receipts, monthly expenditure (as a percentage of the household's monthly SNAP benefit) for whole grain foods in the third month of the intervention period will be compared to the percent of the SNAP benefit during the baseline month (run-in phase). The change in this expenditure amount will be evaluated for intervention participants compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: June Tester, MD MPH, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- UCSF Benioff Children's Hospital Oakland, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Undecided